CLINICAL TRIAL: NCT06904807
Title: A Phase I, Single Ascending and Multiple Ascending Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LIFE-001
Brief Title: A Phase I Study to Evaluate LIFE-001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LifeMine Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIFE-001-1001
Record Dates: First submitted 2025-03-14; First posted 2025-04-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LIFE-001 Single Ascending Dose Cohorts (Experimental): LIFE-001
  Interventions: Drug: LIFE-001
- Placebo Single Ascending Dose Cohorts (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- LIFE-001 Multiple Ascending Dose Cohorts (Experimental): LIFE-001
  Interventions: Drug: LIFE-001 MAD
- Placebo Multiple Ascending Dose Cohorts (Placebo Comparator): Placebo
  Interventions: Drug: Placebo MAD

INTERVENTIONS:
Drug: LIFE-001 — Single dose of LIFE-001 between 10mg and 500mg administered subcutaneously
  Arms: LIFE-001 Single Ascending Dose Cohorts
Drug: Placebo — Single dose of placebo comparator administered subcutaneously
  Arms: Placebo Single Ascending Dose Cohorts
Drug: LIFE-001 MAD — Four doses of LIFE-001 between 50mg and 500mg administered subcutaneously seven days apart
  Arms: LIFE-001 Multiple Ascending Dose Cohorts
Drug: Placebo MAD — Four doses of placebo comparator administered subcutaneously seven days apart
  Arms: Placebo Multiple Ascending Dose Cohorts

SUMMARY:
The goal of this clinical trial is to learn if LIFE-001 is safe and tolerable for healthy adult volunteers.

DETAILED DESCRIPTION:
Participants will attend the site where dosing will be done subcutaneously via direct staff administration and they can only participate in one of the following cohorts:

Single Ascending Dose (SAD) Cohorts 1-7: Screening/baseline period of up to 28 days with a 6-day inpatient say and total duration up to 51 days. Single ascending doses of LIFE-001 between 10mg and 500mg or placebo (Day 1) administered under fasting conditions. Increases will be based on safety and tolerability at each dose level.

Multiple Ascending Dose (MAD) Cohorts 1-5: Screening/baseline period of up to 28 days with two 6-day inpatient says and total duration up to 91 days. Four doses of LIFE-001 between 50mg and 500mg or placebo on Days 1, 8, 15 and 22 administered under fasting conditions.

Exact dose of LIFE-001 for SAD Cohorts 2-7 and MAD will be based on safety, tolerability and pharmacokinetic data from preceding cohorts. After all participants have complete Day 8 (SAD) or Day 29 (MAD), a safety review committee (SRC) will determine if the next dose level cohort will be initiated.

ELIGIBILITY:
Inclusion Criteria:

* Female or male between the ages of 18 and 65 years, inclusive
* Medically healthy (without significant medical issues, e.g. high blood pressure)
* Must provide written informed consent

Exclusion Criteria:

* Ongoing or history of any psychiatric, medical or surgical condition that might jeopardize the participant's safety or interfere with the absorption, distribution or excretion of the study drug
* Any abnormal ECG findings, laboratory value or physical examination findings
* Positive ethanol, drug screen or cotinine test
* Use of systemic prescription medications or over-the-counter (OTC) medication, including multivitamins, and dietary and herbal supplement within 7 days
* Use of any experimental or investigational device within 30 days
* Donation or loss of 500 mL or more of blood within 30 weeks and/or donation of plasma within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | SAD: Predose and Day 1 though Day 22 postdose; MAD: Predose and Day 1 through 56 post initial dose.
  Participant and clinician-reported adverse events

SECONDARY OUTCOMES:
Plasma concentration | SAD: Predose and Day 1 through 22 postdose; MAD: Predose and Day 1 through 56 post initial dose.
  Plasma concentration of LIFE-001
Cmax | SAD: Predose and Day 1 through 22 postdose; MAD: Predose and Day 1 through 56 post initial dose.
  Maximum observed concentration of LIFE-001
Tmax | SAD: Predose and Day 1 through 22 postdose; MAD: Predose and Day 1 through 56 post initial dose.
  Time to maximum observed concentration of LIFE-001

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hall, Principal Investigator — Veritus Research
Locations (1):
- Veritus Research Pty Ltd, Bayswater, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No